CLINICAL TRIAL: NCT01479426
Title: Efficacy and Safety of EFLA400 Korea Red Ginseng Extract on Erectile Dysfunction
Brief Title: A Trial to Evaluate the Efficacy and Safety of EFLA400 Korea Red Ginseng Extract on Sexual Function in Men With Erectile Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Soo-Wan Chae, Clinical Trial Center for Functional Foods, Chonbuk National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: LOTTE-MS-EFLA400
Record Dates: First submitted 2011-11-16; First posted 2011-11-24 (Estimated); Results first posted 2019-09-23 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-08

CONDITIONS: Healthy Subjects(Only Men)
Keywords: Erectile dysfunction; Korean Red Ginseng; IIEF(International Index of Erectile Function); MSHQ(Male Sexual Health Questionnaire,)
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EFLA400(960mg) (Experimental)
  Interventions: Dietary Supplement: EFLA400
- Placebo(960mg) (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: EFLA400 — EFLA400(960mg/day)for 12 weeks
  Other Names: EFLA400 Korean red ginseng
  Arms: EFLA400(960mg)
Dietary Supplement: Placebo — Placebo(960mg/day) for 12 weeks
  Arms: Placebo(960mg)

SUMMARY:
Korea red ginseng has been used in maintaining vitality throughout the globally and metabolism and actions on neurologic, cardiovascular, and endocrinologic system are studied. KRG has been used in various ailment, and to prove its efficacy for erectile dysfunction an international study on contries other than Korean was performed. In the present study, subjects with borderline organic and psychogenic erectile dysfunction will be included. KRG will be give daily, and placebo will be give as control. Outcomes including libido, erection, sexual activity, and sexual satisfaction will be measured.

DETAILED DESCRIPTION:
Among the three main lines of therapy for erectile dysfunction (ED), that is, oral therapy, self-injection therapy and penile prosthesis implantation, the first line therapy is always the first option. Despite the successful advent of sildenafil, the first effective oral agent for ED, further development of new drugs and phytochemical studies of widely known herbal plants are desirable. Furthermore, there seems to be a large population that prefers to use phytotherapies rather than pharmaceutical drugs for their health. Korean red ginseng, a phytotherapy plants, used frequently for ED. Ginseng is one of the most popular herbs in both Eastern and Western countries. It is known as a traditional Asian medicine for stimulation of sexual function and studies have shown the effects of ginseng on relaxation of penile corpus cavernous smooth muscle in many studies. In the present study, the investigators will be determined the real role of Korean red ginseng in the treatment of ED.

ELIGIBILITY:
Inclusion Criteria:

* aged 17-70 years
* IIEF(International Index of Erectile Function)-5 scores ≤ 21 subjects.

Exclusion Criteria:

* they had other neurologic or psychiatric disorder
* significant hepatic or renal function impairment (hepatic enzymes >1.5 times the upper limit of normal and/or serum creatinine >1.8 mg per 100 ml)
* hypertension (>170/110 mm Hg), hypotension (<90/50 mm Hg) or significant cardiovascular disease (unstable angina, coronary artery disease, myocardial infarction or myocardial revascularization).
* Peyronie's disease

Ages: 19 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2010-12; Primary Completion 2011-12 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jong-Kwan Park, MD, Principal Investigator — Chonbuk National University Hospital
Locations (1):
- Clinical Trial Center for Functional Foods; Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea

REFERENCES:
- [Derived] Lee HW, Lee MS, Kim TH, Alraek T, Zaslawski C, Kim JW, Moon DG. Ginseng for erectile dysfunction. Cochrane Database Syst Rev. 2021 Apr 19;4(4):CD012654. doi: 10.1002/14651858.CD012654.pub2. PMID 33871063

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through local advertising and doctor referrals from hospital outpatients and general practice clinics.
Pre-assignment Details: The criteria were an age from 19 to 70 years, IIEF(International Index of Erectile Function)-5 scores ≤ 21 subjects.
Groups:
- EFLA400: EFLA400(2times/day, 2capsules/day, 960mg/day) for 12weeks
  EFLA400: Red Ginseng (90%) and Crataegus pinnatifida Bunge (10%) to high temperature (110 ~ 120 ˚ C) were reacted in the ginsenoside Rg3 increased by alcohol extraction after manufacture.
- Placebo: Placebo(2times/day, 2capsules/day, 960mg/day) for 12weeks
  Placebo : Amount and calorie of placebo are same with EFLA400
Period: Overall Study
Arm/Group | EFLA400 | Placebo
Started | 40 | 40
Completed | 36 | 37
Not Completed | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EFLA400(960mg) | Placebo(960mg) | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 40 | 80
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.13 (6.65) | 59.70 (7.59) | 59.91 (7.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 40 | 40 | 80
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: Changes in EF(Erectile Function) Domain
Description: EF(erectile function, score 0-20) domain was measured in study visit 1(0 week) and visit 3(12 week).
  The original index consists of 4 Questions. Individual question response is assigned a score of between 0 (worst) to 5 (best) and summed to form a score ranging from 0 (worst) to 20 (best).
Time Frame: 12 weeks
Population: per protocol analysis
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- EFLA400: Oral intake EFLA400(960mg/day) for 12weeks.
- Placebo: Oral intake placebo(960mg/day) for 12weeks.
Arm/Group | EFLA400 | Placebo
Number analyzed (Participants) | 36 | 37
Scores on a scale
  Pre | 11.53 (4.33) | 12.89 (4.19)
  Post | 14.56 (4.92) | 16.46 (5.16)

2. Secondary Outcome: Changes in MSHQ (Male Sexual Health Questionnaire)
Description: MSHQ(Male Sexual Health Questionnaire) was measured in study visit 1(0 week) and visit 3(12 week).
  The total MSHQ score (25 questions) ranges from 17-130, with higher scores indicating greater sexual function.
Time Frame: 12 weeks
Population: per protocol analysis
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | EFLA400 | Placebo
Number analyzed (Participants) | 36 | 37
Scores on a scale
  Pre | 70.28 (12.98) | 71.62 (14.80)
  Post | 82.22 (17.34) | 83.81 (19.19)

3. Secondary Outcome: GEAQ (Global Efficacy Assessment Question)
Time Frame: after 12weeks of consumption
Reporting Status: Not Posted

4. Secondary Outcome: Changes in Uroflowmetry(Max Flow Rate)
Description: uroflowmetry(max flow rate) was measured in study visit 1(0 week) and visit 3(12 week).
Time Frame: 12 weeks
Population: per protocol analysis
Measure: Mean (Standard Deviation); unit: m/sec
Arm/Group | EFLA400 | Placebo
Number analyzed (Participants) | 36 | 37
m/sec
  Pre | 19.65 (9.48) | 17.64 (6.47)
  Post | 20.63 (8.96) | 20.95 (9.46)

5. Secondary Outcome: Changes in IIEF(International Index of Erectile Function)-Total Domain
Description: IIEF(International Index of Erectile Function)-total domain(score range: 5-75) was measured in study visit 1(0 week) and visit 3(12 week).
  IIEF includes 15 questions and addresses the 5 sub-domains of Erectile function, Intercourse satisfaction, Orgasm function, Sexual desire, and Overall satisfaction.
  The IIEF-total domain is the sum of sub-domains. Lower scores indicate severe erectile dysfunction, while higher scores indicate less erectile dysfunction.
Time Frame: 12 weeks
Population: per protocol analysis
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | EFLA400 | Placebo
Number analyzed (Participants) | 36 | 37
Scores on a scale
  Pre | 37.83 (10.89) | 41.00 (10.30)
  Post | 47.11 (12.04) | 50.41 (12.58)

ADVERSE EVENTS:
Description: Serious and/or other [non-serious] adverse events were not collected/assessed
Arm/Group | EFLA400(960mg) | Placebo(960mg)
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No